CLINICAL TRIAL: NCT04581317
Title: Connecting Seniors to Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: U.S. Administration for Community Living (Unknown)
Responsible Party: Principal Investigator, Jessica Lee, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-20-0857
Record Dates: First submitted 2020-10-02; First posted 2020-10-09 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Dementia
Keywords: nutrition; virtual assistant device; frailty; social determinants of health
MeSH Terms: conditions — Dementia; Frailty | interventions — Meals

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1 (meals only) (Experimental): Participants will receive meals delivered to them by the Meals oN wheels(MOW) program for 6 weeks.MOW will once a week deliver in-person enough frozen meals to cover lunch for 5 days and breakfast for 7 days. Study staff will call the participants twice a week to ask 5 questions about their health, mood, and meal consumption.At the end of the 6 weeks, a study team member will make an in-person visit to the participants' homes to measure Fried Frailty Phenotype(FFP), MHS, CES-D, MOCA, Activities of Daily Living (ADL)/Instrumental activities of daily living(IADL)s, NSI, and ZCBI. Caregivers will not receive meals during this first phase as the focus is on the nutritional status of the cognitively impaired older adult.
  Interventions: Other: meals
- Phase 2 (Meals + Amazon Echo Show 8 (AES 8) basic usage) (Experimental): Participants will have meals delivered and the AES device installed for basic usage
  Interventions: Other: meals; Other: AES 8 basic usage
- Phase 3 (meals + AES 8 advanced ) (Experimental): Participants will have meals delivered and the AES device installed for advanced usage
  Interventions: Other: meals; Other: AES 8 advanced usage

INTERVENTIONS:
Other: meals — Participants will receive meals delivered to them by the Meals oN wheels(MOW) program for 6 weeks.
Other: AES 8 basic usage — For the second 6 weeks, participants will continue to have meal deliveries and will now have the AES 8 device which can be used by the cognitively impaired participant and their caregiver. AES 8 devices will be installed in participant's homes by the study team and participants will be given basic instructions on using the device as well as a one-page handout that will include instructions on how to use and maintain privacy with their device. The study staff will continue to call twice a week to ask the 5 questions. At the end of the 6 weeks, a study team member will make an in-person visit to the participants' homes to measure FFP, MHS, CES-D, MOCA, ADL/IADLs, NSI, ZCBI, and TAM.
  Arms: Phase 2 (Meals + Amazon Echo Show 8 (AES 8) basic usage)
Other: AES 8 advanced usage — In the third 6 weeks, the participants will continue to have meal deliveries and the AES 8 will be upgraded to provide an active intervention by asking the twice a week 5 questions through the device. The questions should be answered by the cognitively impaired older adult using the device, though the caregiver can still use the device for other basic services. The participant will be able to answer the questions verbally or by touch screen options displayed on the device.At the end of the 6 weeks, a study team member will make an in-person visit to the participants' homes to measure FFP, MHS, CES-D, MOCA, ADL/IADLs, NSI, ZCBI, and TAM.
  Arms: Phase 3 (meals + AES 8 advanced )

SUMMARY:
The purpose of this study is to assess the feasibility of implementing the virtual assistant devices into the daily routine of participants and their caregivers,to measure social determinants of health,depression,cognitive impairment,nutritional and functional status in the cognitively impaired participants

ELIGIBILITY:
Inclusion Criteria:

* cognitive impairment as reported in the Mental Health Screening/Assessment section on the Interfaith Ministries of Greater Houston's Meals on Wheels Program (IMGH MOW) intake form
* are on the IMGH MOW waiting list
* medically stable

Exclusion Criteria:

* do not have cognitive impairment
* have a pre-diagnosed terminal illness
* unable to ambulate, and/or are unable to use their upper extremities.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by the technology acceptance measure (TAM) | 12 weeks from baseline
  The TAM has 4 questions each one with five answer choices ranging form Strongly Agree to Strongly Disagree
Feasibility as measured by the technology acceptance measure (TAM) | 18 weeks from baseline
  The TAM has 4 questions each one with five answer choices ranging form Strongly Agree to Strongly Disagree

SECONDARY OUTCOMES:
Change in social determinants of health as measured by the the Mental Health Screening/Assessment (MHS) | Baseline,18 weeks
Change in Depression as measured by the Center for Epidemiologic Studies Depression Scale (CES-D) | Baseline,18 weeks
  The scale consists of 20 questions and each is scored from 0-4,a higher number indicating more depression
Change in cognitive impairment as measured by the Montreal Cognitive Assessment (MOCA) | Baseline,18 weeks
  Total score on the Montreal Cognitive Assessment (MoCA) range from 0 to 30, with a higher score indicating a better outcome.
Change in nutritional status as measured by the Nutrition Screening Initiative (NSI) | Baseline,18 weeks
Change in Caregiver burden as measured by the Zarit Caregiver Burden Interview (ZCBI) | Baseline,18 weeks
  The ZCBI has 22 questions with a score ranging from 0-88, a higher score indicating more burden

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Lee, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nunez M, Patel P, Ulin L, Kian L, Cominsky M, Burnett J, Lee JL. Feasibility and Usage of a Virtual Assistant Device in Cognitively Impaired Homebound Older Adults. J Appl Gerontol. 2025 Oct;44(10):1651-1660. doi: 10.1177/07334648251314284. Epub 2025 Jan 10. PMID 39792590